CLINICAL TRIAL: NCT06714448
Title: Post Authorization Safety Study Assessing the Effectiveness of Risk Minimization Measures Related to Depakine® (Sodium Valproate) in Saudi Arabia
Brief Title: A Study of the Effectiveness of Risk Minimization Measures Related to Depakine® (Sodium Valproate) in Saudi Arabia
Acronym: DEPAKINE PASS
Status: Active, not recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS18507; U1111-1310-4851 (Registry Identifier: WHO ICTRP)
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Epilepsy; Seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Valproic Acid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sodium valporate: Participants are healthcare professionals completing a survey regarding women of childbearing potential using sodium valporate, prescribe or dispense the treatment
  Interventions: Drug: Sodium valporate

INTERVENTIONS:
Drug: Sodium valporate — This study will not administer any treatment, only observe the treatment as prescribed in real-world clinical practices.
  Other Names: Depakine®

SUMMARY:
A cross-sectional, national, multicenter, survey-based study to assess the effectiveness of Risk Minimization Measures related to Depakine® (sodium valproate) in Saudi Arabia. The end of study is defined as the end of the data collection period. No intervention will be administered, and no study related visits are required.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals working only in Saudi Arabia AND
* Prescribers of Depakine® (sodium valiporate) at least once in the six months leading up to survey completion OR
* Obstetricians/Gynecologists who consulted at least one women of childbearing potential treated with Depakine® (sodium valproate) in the six months leading up to survey completion OR
* Pharmacists who have dispensed Depakine® (sodium valproate) in the six months leading up to survey completion

Exclusion Criteria:

* Healthcare professionals who may have conflicts of interest with the survey (i.e. employed by regulatory bodies or pharmaceutical companies)
* Healthcare professionals (or with a relative) involved in valproate-related lawsuits or associations for victims of valproate syndrome
* Healthcare professionals who are not prescribing Depakine® (sodium valproate), except for obstetricians/gynecologists (who do not prescribe Depakine® [sodium valproate])
* Healthcare professionals having started to prescribe or dispense Depakine® (sodium valproate) earlier than six months before survey completion

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: In this survey-based study, the data will be collected from each healthcare professional participant in Saudi Arabia once at a certain time. However, the study will take 7 months, from 30 November 2024 to 30 May 2025, to collect the required number of responses.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2025-11-27 (Estimated); Study Completion 2025-11-27 (Estimated)

PRIMARY OUTCOMES:
Percentage of healthcare professionals who received and read the educational materials | 7 months
Healthcare professionals' knowledge score | 7 months
  Knowledge score is calculated as the proportion of correct responses among all questions related to knowledge
Healthcare professionals' behavior score | 7 months
  Behavior score is calculated as the proportion of correct responses among all questions related to behavior

CONTACTS AND LOCATIONS:
Locations (1):
- Sanofi-Aventis, Chilly-Mazarin, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org